CLINICAL TRIAL: NCT00582075
Title: Phase II Study of Gamma Knife Radiosurgery and Temozolomide (Temodar) for Newly Diagnosed Brain Metastases
Brief Title: Phase II Study of Gamma Knife Radiosurgery and Temozolomide for Brain Metastases
Acronym: RAD0102
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Integrated Therapeutics Group (Industry)
Responsible Party: Principal Investigator, John Fiveash, MD, Professor and Vice Chair, University of Alabama at Birmingham Department of Radiation Oncology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F020522015
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Cancer; Brain Metastases
Keywords: Cancer; Brain metastases; Gamma Knife Radiosurgery; Temodar; Temozolomide
MeSH Terms: conditions — Neoplasms; Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiosurgery 15-24 Gy + Adjuvant Temozolomide (Experimental)
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide — TMZ 200mg/m2 days 1-5 repeat q28 days. Patients who have received prior chemotherapy will receive 150 mg/m2 days 1-5
  Other Names: Temodar

SUMMARY:
The protocol is designed to determine the efficacy of temozolomide in preventing the development of new brain metastases within the first year in patients undergoing stereotactic radiation for newly diagnosed brain metastases.

DETAILED DESCRIPTION:
This is a phase II study. The primary endpoint is the proportion of patients with newly developed metastases who develop new brain metastases within the first year of undergoing stereotactic radiation combined with the administration of temozolamide within the first year post treatment. Retrospective and prospective studies suggest that 50- 60% of long-term survivors develop new brain metastases. Since it is important to observe all patients recruited for a minimum of a year to measure the primary outcome, traditional phase 2 designs such as Simon's two stage optimal design or the mini-max design are not practical in this case. Survival and QOL are secondary end points. QOL will be measured using the Functional Assessment of Cancer Therapy (FACT -BR). It will be administered at baseline, at week four and every three months for 24 months.

This protocol includes radiosurgery with standard radiation doses (15-24 Gy based upon RTOG 9005). Patient may be registered after radiosurgery as long as Temodar is started within two weeks of radiosurgery.

Beginning within two weeks after radiosurgery: TMZ 200mg/m2 days 1-5 repeat q28 days. Patients who have received prior chemotherapy will receive 150 mg/m2 days 1-5.

Temozolomide is continued until there is disease progression defined by systemic progression or new metastases. If lesion treated with radiosurgery progresses in the absence of new CNS tumors or systemic progression, then TMZ will continue. Temozolomide is discontinued for systemic progression requiring other systemic chemotherapy.

Palliative radiation may be administered to non-CNS sites during protocol treatment, but additional systemic chemotherapy will not be administered until patients progress systemically or until new metastases develop.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have history of histologically confirmed malignancy. Brain biopsy is not required unless diagnosis is judged to be in doubt by the treating physician.
* Newly diagnosed brain metastases (four or fewer by thin slice post-contrast MRI).
* ECOG performance status of less than or equal to 2 for patients with no prior chemotherapy, and less than or equal to 1 for patients with prior chemotherapy.
* Age greater than 18
* Life expectancy greater than 12 weeks
* Subjects given written informed consent
* Adequate hematologic, renal and liver function as demonstrated by laboratory values performed within 14 days, inclusive, prior to administration of study drug:

  * Absolute neutrophil count (ANC) >= 1500/mm3
  * Platelet count >= 100,000/mm3
  * Hemoglobin >= 9 g/dL
  * BUN and serum creatinine <= 1.5 times upper limit of laboratory normal
  * Total and direct bilirubin <= 2 times upper limit of laboratory normal or in the presence of documented liver metastases, total and direct bilirubin <=5 times upper limit of normal
  * SGOT and SGPT <= 2 times upper limit of laboratory normal or in the presence of documented liver metastases, SGOT and SGPT <=5 times upper limit of normal
  * Alkaline phosphatase <= 2 times upper limit of laboratory normal or in the presence of documented liver metastases, alkaline phosphatase of <= 5 times upper limit of normal

Exclusion Criteria:

* Patients with small cell lung cancer and lymphoma are ineligible.
* More than four metastases by thin slice MRI. Note that if a diagnostic study prior to radiosurgery demonstrates only four tumors but the gamma knife treatment-planning scan reveals greater than four tumors, the patients will still be eligible for the protocol if all tumors can be treated with radiosurgery.
* Chemotherapy within four weeks prior to study drug administration
* Patients, who in the opinion of the treating medical oncologist, require immediate cytotoxic chemotherapy other than the study drug. Allowed medications include antihormonal agents (i.e., Tamoxifen), herceptin and bisphosphonates.
* Radiation therapy to greater than or equal to 50% of the bone marrow. Completion of radiation therapy less than 4 weeks prior to study drug administration for radiotherapy to >= 15% of bone marrow and less than 2 weeks prior for radiotherapy to < 15% of bone marrow.
* Insufficient recovery from all active toxicities of prior therapies
* Subjects who are poor medical risks because of non-malignant systemic disease
* Frequent vomiting or medical condition that could interfere with oral medication intake (e.g., partial bowel obstruction).
* Previous or concurrent malignancies at other sites, or treatment for malignancy at the site within 5 years of study start with the exception of surgically cured carcinoma in-situ of the cervix and basal or squamous cell carcinoma of the skin.
* Known HIV positively or AIDS-related illness.
* Pregnant or nursing women.
* Women of childbearing potential who are not using an effective method of contraception. Women of childbearing potential must have a negative serum pregnancy test 24 hours prior to administration of study drug and be practicing medically approved contraceptive precautions.
* Men who are not advised to use an effective method of contraception.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-07; Primary Completion 2008-10 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fiveash, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] DeAngelis LM, Delattre JY, Posner JB. Radiation-induced dementia in patients cured of brain metastases. Neurology. 1989 Jun;39(6):789-96. doi: 10.1212/wnl.39.6.789. PMID 2725874
- [Background] Pirzkall A, Debus J, Lohr F, Fuss M, Rhein B, Engenhart-Cabillic R, Wannenmacher M. Radiosurgery alone or in combination with whole-brain radiotherapy for brain metastases. J Clin Oncol. 1998 Nov;16(11):3563-9. doi: 10.1200/JCO.1998.16.11.3563. PMID 9817276
- [Background] Sneed PK, Lamborn KR, Forstner JM, McDermott MW, Chang S, Park E, Gutin PH, Phillips TL, Wara WM, Larson DA. Radiosurgery for brain metastases: is whole brain radiotherapy necessary? Int J Radiat Oncol Biol Phys. 1999 Feb 1;43(3):549-58. doi: 10.1016/s0360-3016(98)00447-7. PMID 10078636
- [Background] Patchell RA, Tibbs PA, Regine WF, Dempsey RJ, Mohiuddin M, Kryscio RJ, Markesbery WR, Foon KA, Young B. Postoperative radiotherapy in the treatment of single metastases to the brain: a randomized trial. JAMA. 1998 Nov 4;280(17):1485-9. doi: 10.1001/jama.280.17.1485. PMID 9809728
- [Background] Stevens MF, Hickman JA, Stone R, Gibson NW, Baig GU, Lunt E, Newton CG. Antitumor imidazotetrazines. 1. Synthesis and chemistry of 8-carbamoyl-3-(2-chloroethyl)imidazo[5,1-d]-1,2,3,5-tetrazin-4(3 H)-one , a novel broad-spectrum antitumor agent. J Med Chem. 1984 Feb;27(2):196-201. doi: 10.1021/jm00368a016. PMID 6694168
- [Background] Tsang LL, Quarterman CP, Gescher A, Slack JA. Comparison of the cytotoxicity in vitro of temozolomide and dacarbazine, prodrugs of 3-methyl-(triazen-1-yl)imidazole-4-carboxamide. Cancer Chemother Pharmacol. 1991;27(5):342-6. doi: 10.1007/BF00688855. PMID 1998993
- [Background] Bull VL, Tisdale MJ. Antitumour imidazotetrazines--XVI. Macromolecular alkylation by 3-substituted imidazotetrazinones. Biochem Pharmacol. 1987 Oct 1;36(19):3215-20. doi: 10.1016/0006-2952(87)90636-8. PMID 2444229
- [Background] Tisdale MJ. Antitumour imidazotetrazines--XVIII. Modification of the level of 5-methylcytosine in DNA by 3-substituted imidazotetrazinones. Biochem Pharmacol. 1989 Apr 1;38(7):1097-101. doi: 10.1016/0006-2952(89)90254-2. PMID 2706009
- [Background] Tsang LL, Farmer PB, Gescher A, Slack JA. Characterisation of urinary metabolites of temozolomide in humans and mice and evaluation of their cytotoxicity. Cancer Chemother Pharmacol. 1990;26(6):429-36. doi: 10.1007/BF02994094. PMID 2225314
- [Background] Clark AS, Stevens MF, Sansom CE, Schwalbe CH. Anti-tumour imidazotetrazines. Part XXI. Mitozolomide and temozolomide: probes for the major groove of DNA. Anticancer Drug Des. 1990 Feb;5(1):63-8. PMID 2317259
- [Background] Stevens MF, Hickman JA, Langdon SP, Chubb D, Vickers L, Stone R, Baig G, Goddard C, Gibson NW, Slack JA, et al. Antitumor activity and pharmacokinetics in mice of 8-carbamoyl-3-methyl-imidazo[5,1-d]-1,2,3,5-tetrazin-4(3H)-one (CCRG 81045; M & B 39831), a novel drug with potential as an alternative to dacarbazine. Cancer Res. 1987 Nov 15;47(22):5846-52. PMID 3664486
- [Background] Gibson NW, Hickman JA, Erickson LC. DNA cross-linking and cytotoxicity in normal and transformed human cells treated in vitro with 8-carbamoyl-3-(2-chloroethyl)imidazo[5,1-d] -1,2,3,5-tetrazin-4(3H)-one. Cancer Res. 1984 May;44(5):1772-5. PMID 6713381
- [Background] Hartley JA, Gibson NW, Kohn KW, Mattes WB. DNA sequence selectivity of guanine-N7 alkylation by three antitumor chloroethylating agents. Cancer Res. 1986 Apr;46(4 Pt 2):1943-7. PMID 3004713
- [Background] SN92384: SCH 52365: Pharmacokinetics of SCH 52365 in Rats Following a Single Oral Gavage or Intravenous Dose. Schering-Plough Research Institute
- [Background] SN92385: SCH 52365: Pharmacokinetics of SCH 52365 in Beagle Dogs Following a Single Oral Gavage or a Single Intravenous Cross-Over Study. Schering Plough Research Institute
- [Background] SN92131: Single-Cycle Oral Toxicity Study of SCH 52365 in Rats. Schering Plough Research Institute.
- [Background] SN93092: Single-Cycle Oral Toxicity Study with Lower Doses of SCH 52365 in Rats. Schering-Plough Research Institute
- [Background] SN92133: Three-Cycle Oral Toxicity Study of SCH 52365 in Rats. Schering Plough Research Institute.
- [Background] SN92132: Single-Cycle Oral Toxicity Study of SCH 52365 in Dogs. Schering-Plough Research Institute
- [Background] SN93093: Single-Cycle Oral Toxicity Study with Lower Doses of SCH 52365 in Dogs. Schering-Plough Research Institute
- [Background] SN92134: Three-Cycle Oral Toxicity Study of SCH 52365 in Dogs. Schering-Plough Research Institute
- [Background] SN92380: SCH 52365: Mass Balance and Excretion of 14C-SCH 52365 Following a Single Intravenous or Oral Dose in Male Rats. Schering-Plough Research Institute
- [Background] SN92383: SCH 52365: Absorption, Distribution and Metabolism of 14C SCH 52365 Following a Single Oral Dose in Male Rats. Schering-Plough Research Institute
- [Background] SN92381: SCH 52365: Absorption, Metabolism, Excretion, and Pharmacokinetics of 14C-SCH 52365 Following a Single Oral or Intravenous Dose in the Male Rat. Schering-Plough Research Institute
- [Background] SN92382: SCH 52365: Absorption, Metabolism, Excretion, and Pharmacokinetics of 14C-SCH 52365 Following a Single Oral And Intravenous Dose in the Male Dog. Schering-Plough Research Institute
- [Background] Patel M, McCully C, Godwin K, Balis FM. Plasma and cerebrospinal fluid pharmacokinetics of intravenous temozolomide in non-human primates. J Neurooncol. 2003 Feb;61(3):203-7. doi: 10.1023/a:1022592913323. PMID 12675312
- [Background] Newlands ES, Blackledge GR, Slack JA, Rustin GJ, Smith DB, Stuart NS, Quarterman CP, Hoffman R, Stevens MF, Brampton MH, et al. Phase I trial of temozolomide (CCRG 81045: M&B 39831: NSC 362856). Br J Cancer. 1992 Feb;65(2):287-91. doi: 10.1038/bjc.1992.57. PMID 1739631
- [Background] O'Reilly SM, Newlands ES, Stevens MFG, Brampton MH, Slack JA et al: Temozolomide (CCRG 81045; M&B 39831; NSC 362856): a new oral cytotoxic agent with activity against melanoma, mycosis fungoides and high-grade glioma. Proc. AACR. 1992; 33: A1267
- [Background] O'Reilly SM, Newlands ES, Glaser MG, Brampton M, Rice-Edwards JM, Illingworth RD, Richards PG, Kennard C, Colquhoun IR, Lewis P, et al. Temozolomide: a new oral cytotoxic chemotherapeutic agent with promising activity against primary brain tumours. Eur J Cancer. 1993;29A(7):940-2. doi: 10.1016/s0959-8049(05)80198-4. PMID 8499146
- [Background] Data on file at the Cancer Research Campaign Data Center. Phase II trial of temozolomide in high-grade glioma. Schering-Plough Research Institute. Study No. H93-090-50).
- [Background] Data on file at the Cancer Research Campaign Data Center. Phase II trial of temozolomide in advanced malignant melanoma. Schering-Plough Research Institute. Study No. H93 088-50
- [Background] Bleehen NM, Newlands ES, Lee SM, Thatcher N, Selby P, Calvert AH, Rustin GJ, Brampton M, Stevens MF. Cancer Research Campaign phase II trial of temozolomide in metastatic melanoma. J Clin Oncol. 1995 Apr;13(4):910-3. doi: 10.1200/JCO.1995.13.4.910. PMID 7707118
- [Background] Data on file at the Cancer Research Campaign Data Center. Phase II trial of temozolomide in low-grade non-Hodgkin's lymphoma. Schering-Plough Research Institute. Study No. H93-089-50).
- [Background] Woll PJ, Crowther D, Johnson PW, Soukop M, Harper PG, Harris M, Brampton MH, Newlands ES. Phase II trial of temozolomide in low-grade non-Hodgkin's lymphoma. Br J Cancer. 1995 Jul;72(1):183-4. doi: 10.1038/bjc.1995.299. PMID 7599050
- [Background] Data on file at Schering-Plough Research Institute (I93-114-01).
- [Background] Brada M, Moore S, Judson I, Batra VJ, Quartey P, Dugan M: A Phase I study of SCH 52365 (temozolomide) in adult patients with advanced cancer. Proc. ASCO. 1995; 14:1521
- [Background] Data on file at Schering-Plough Research Institute (C94-022-01).
- [Background] Hammond LA, Eckardt JR, Baker SD, Eckhardt SG, Dugan M, Forral K, Reidenberg P, Statkevich P, Weiss GR, Rinaldi DA, Von Hoff DD, Rowinsky EK. Phase I and pharmacokinetic study of temozolomide on a daily-for-5-days schedule in patients with advanced solid malignancies. J Clin Oncol. 1999 Aug;17(8):2604-13. doi: 10.1200/JCO.1999.17.8.2604. PMID 10561328
- [Background] Yung A, Levin VA, Albright R, Olson J, Fredericks R, Fink K, Prados M, Brada M, Spence A, Brunner J, Yue N, Dugan MH, Zaknoen S. Temodal Brain Tumor Group: Randomized trial of temodal (TEM) vs. procarbazine (PCB) in glioblastoma multi-forme (GBM) at first relapse [abstract]. Proceedings of the American Society of Clinical Oncology. 1999; 18:139a.
- [Background] Christodoulou C, Bafaloukos D, Kosmidis P, Samantas E, Bamias A, Papakostas P, Karabelis A, Bacoyiannis C, Skarlos DV; Hellenic Cooperative Oncology Group. Phase II study of temozolomide in heavily pretreated cancer patients with brain metastases. Ann Oncol. 2001 Feb;12(2):249-54. doi: 10.1023/a:1008354323167. PMID 11300333
- [Background] Paraskevaidis E, Antonadou D, Sarris G, Kolliarakis N, Economou I, Karageirgus P, Throuvalas N. A Phase II randomized trial of synchronous radiotherapy with temozolomide in brain metastases. Metaxas Cancer Hospital, Pireus, Greece
- [Result] Abrey JD, Olson DY, Boutros M, Mack A, Rodavitch JJ, Raizer MG. A Phase II Study of Temozolomide for Recurrent Brain Metastases. Malkin; Memorial Sloan-Kettering Cancer Center, New York, NY. Abstract 643

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiosurgery 15-24 Gy + Adjuvant Temozolomide: Patients with newly diagnosed brain mets treated with radiosurgery.
Period: Overall Study
Arm/Group | Radiosurgery 15-24 Gy + Adjuvant Temozolomide
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiosurgery 15-24 Gy + Adjuvant Temozolomide
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 56 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Distant Brain Failure (DBF) at One Year
Description: Patients developing distant brain failure (DBF) at one year. An approximation method was used to arrive at the reported percentage.
Time Frame: 1 years
Measure: Number; unit: percentage of participants
Arm/Group | Radiosurgery 15-24 Gy + Adjuvant Temozolomide
Number analyzed (Participants) | 25
percentage of participants | 37

2. Secondary Outcome: Overall Survival
Time Frame: 2 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Radiosurgery 15-24 Gy + Adjuvant Temozolomide
Number analyzed (Participants) | 25
weeks | 31 [11 to 104]

ADVERSE EVENTS:
Arm/Group | Radiosurgery 15-24 Gy + Adjuvant Temozolomide
Serious Adverse Events (participants affected / at risk) | 15/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiosurgery 15-24 Gy + Adjuvant Temozolomide (N=25)
DVT (Vascular disorders) | 3
Broken Hip (Musculoskeletal and connective tissue disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Nausea and Vomiting (Gastrointestinal disorders) | 1
Death (Cardiac disorders) | 1 — Death at home of apparent heart attack. No autopsy.
Seizures (Nervous system disorders) | 1
Surgical Revision of Necrotic Tissue (Surgical and medical procedures) | 2
Hemorrhage (GI) (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Altered Mental Status (Nervous system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiosurgery 15-24 Gy + Adjuvant Temozolomide (N=25)
Hyperglycemia (Metabolism and nutrition disorders) | 16
Lymphopenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Anemia (Blood and lymphatic system disorders) | 11
Hypoalbuminemia (Investigations) | 12
Decreased White Blood Cell Count (Blood and lymphatic system disorders) | 10
Hyperkalemia (Investigations) | 2
Constipation (Gastrointestinal disorders) | 8
Increased ALT (Investigations) | 8
Fever (General disorders) | 3
Hyponatremia (Investigations) | 5
Hypocalcemia (Investigations) | 3
Confusion (Nervous system disorders) | 4
Fatigue (General disorders) | 11
Hypoglycemia (Investigations) | 2
Nausea (Gastrointestinal disorders) | 10
Hypokalemia (Investigations) | 2
Hypernatremia (Investigations) | 2
Increased Bilirubin (Investigations) | 3
Headache (Nervous system disorders) | 10
Diarrhea (Gastrointestinal disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Vision Alteration (Nervous system disorders) | 4
Dizziness (General disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Ataxia (Nervous system disorders) | 2
Increased GGT (Investigations) | 2
Decreased ANC (Blood and lymphatic system disorders) | 4
Increased AST (Investigations) | 3
Weakness (General disorders) | 2
Vertigo (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 3
Neuropathy - Motor (Nervous system disorders) | 2
Radionecrosis (Injury, poisoning and procedural complications) | 2
Anorexia (General disorders) | 2
Syncope (Nervous system disorders) | 2
Neuropathy - Sensory (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes